CLINICAL TRIAL: NCT02477943
Title: Objective Brain Function Assessment of mTBI From Initial Injury to Rehabilitation and Treatment Optimization in College Athletes
Brief Title: Objective Brain Function Assessment of mTBI/Concussion in College Athletes
Acronym: AheadCAS
Status: Completed | Type: Observational
Sponsor: BrainScope Company, Inc. (Industry)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 14-Ahead
Record Dates: First submitted 2015-06-15; First posted 2015-06-23 (Estimated); Last update posted 2019-05-23 (Actual); Status verified 2019-05

CONDITIONS: Brain Injuries, Traumatic; Concussion, Mild; Concussion, Brain; Concussion, Intermediate; Concussion, Severe
Keywords: Concussion; Mild Traumatic Brain Injury; Sport Related Concussion
MeSH Terms: conditions — Brain Injuries, Traumatic; Brain Concussion | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Injured and Matched Control Subject Pool: Injured subjects consist of athletes who are head injured and meet the inclusion/exclusion criteria. Injured subjects will be tested within 72 hours (3 days) of injury and at specified time points post injury. Matched control subjects will be tested at the same time intervals as the injured subject. BrainScope Battery will be performed at each time point and consists of the following components: brain electrical activity (EEG), neurocognitive performance assessment, balance/sway measurement, and clinical symptoms/assessments. In addition, a subset of injured and matched control subjects will receive advanced MRI/DTI neuroimaging at time of injury and following RTP.
  Interventions: Device: BrainScope Ahead 200iD; Device: Advanced MRI Neuroimaging
- Pre-Season and Post-Season Subject Pool: This subject pool will consist of uninjured (not head injured) contact and non-contact athletes and will be tested at two time points - pre-season and post-season. These subjects will perform the same BrainScope Battery as the injured and matched control subjects at each time points.
  Interventions: Device: BrainScope Ahead 200iD

INTERVENTIONS:
Device: BrainScope Ahead 200iD — The BrainScope Battery evaluation will consist of 4 tests to aid in the assessment of concussion: History, Physical, signs and symptoms (SAC, SCAT3), Electrophysiological Function; Neurocognitive Performance Assessment and a balance/sway measurement. BrainScope Ahead 200iD device will be used to perform EEG.
Device: Advanced MRI Neuroimaging — Diffusion tensor imaging (DTI) is a magnetic resonance imaging technique that enables the measurement of the restricted diffusion of water in tissue in order to produce neural tract images instead of using this data solely for the purpose of assigning contrast or colors to pixels in a cross sectional image.
  Other Names: Magnetic Resonance Imaging; Diffusion Tension Imaging
  Groups: Injured and Matched Control Subject Pool

SUMMARY:
This study (Part 1) is designed to build a database including EEG, neurocognitive performance, clinical symptoms, history and other relevant data, which will be used to derive a multimodal EEG based algorithm for the identification of concussion and tracking of recovery. In addition, neuroimaging will be conducted at time of injury and following Return to Play (RTP).

DETAILED DESCRIPTION:
Injured/concussed subjects will be studied at time of injury, and at 3 follow-up time points following injury. Matched controls will be tested following the same schedule as the injured athletes. In addition, the study will include an additional pool of contact and non-contact athletes who are not head injured and will be assessed prior to the season and then after the season has ended. This data will be used to populate a database for the purpose of deriving a multimodal concussion index.

ELIGIBILITY:
Inclusion Criteria:

* Concussion-Injury subjects will be defined as follows: Any player who, based on independent clinical impression, is suspected of having suffered a concussion of any severity level, and on whom a routine clinical examination for concussion or head injury would have been conducted prior to implementation of this research protocol according to current standard practice.

  1. If loss of consciousness, total duration less than <20 minutes
  2. No evidence of abnormality visible on Computerized Tomography (CT) of the head related to the traumatic event (Note: neuroimaging is not required for enrollment)
  3. No hospital admission due to either head injury or collateral injuries for >24 hours.
  4. GCS is between 13-15.

Exclusion Criteria:

1. Evidence of illicit drug usage
2. Do not speak or read English
3. Current CNS active prescription medications, with the exception of medications being taken for the treatment of Attention Deficit Disorder (ADD)
4. Skull abnormalities, e.g. metal plate
5. History of brain surgery or neurological disease.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Approximately 450 male and female student-athletes from participating universities or colleges will be invited to participate.
Sampling Method: Non-Probability Sample
Enrollment: 520 (Actual)
Dates: Start 2015-08-08 (Actual); Primary Completion 2017-02-20 (Actual); Study Completion 2017-07-31 (Actual)

PRIMARY OUTCOMES:
Algorithm for Likelihood of being concussed | 6 months for data acquisition, with each patient studied from time of injury to 45 days after RTP
  Create a database of brain electrical activity (EEG) and clinical information collected from athletes who sustain a concussion during organized sports.

SECONDARY OUTCOMES:
Advanced Neuroimaging in concussion | 6 months for data acquisition, with each patient studied from time of injury to 45 days after RTP
  Exploration of changes in functional neuroimaging which occur with concussion and change in these measures over time.

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Prichep, Ph.D., Study Director — BrainScope Company, Inc.
Locations (11):
- United States (11):
  - University of Arkansas, Fayetteville, Arkansas
  - University of Connecticut, Storrs, Connecticut
  - University of South Florida, Tampa, Florida
  - Michigan State University, East Lansing, Michigan
  - University of New Mexico, Albuquerque, New Mexico
  - University of Rochester Medical Center, Rochester, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - University of South Carolina, Columbia, South Carolina
  - University of Texas - Austin, Austin, Texas
  - Baylor College of Medicine, Houston, Texas
  - Houston Methodist Hospital, Houston, Texas

REFERENCES:
- [Derived] Covassin T, McGowan AL, Bretzin AC, Anderson M, Petit KM, Savage JL, Katie SL, Elbin RJ, Pontifex MB. Preliminary investigation of a multimodal enhanced brain function index among high school and collegiate concussed male and female athletes. Phys Sportsmed. 2020 Nov;48(4):442-449. doi: 10.1080/00913847.2020.1745717. Epub 2020 Mar 31. PMID 32228157